CLINICAL TRIAL: NCT03076749
Title: Designing Predictive Models for Betalactam Allergy Using the Drug Allergy and Hypersensitivity Database®
Brief Title: Predictive Models for Betalactam Allergy
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8927; 2012-A00182-41 (Other: Agence Francaise de securité sanitaire des produits de santé)
Record Dates: First submitted 2016-09-09; First posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2012-02

CONDITIONS: Drug Hypersensitivity
Keywords: Betalactam; Decision tree; Drug hypersensitivity; Logistic regression; Predictive modelling
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Creating models for the diagnosis of BL allergy

SUMMARY:
Background: ß-lactam (BL) antibiotics represent the main cause of allergic reactions to drugs, inducing both immediate and non-immediate reactions. The diagnosis is well established, usually based upon skin tests and drug provocation tests, but cumbersome.

Objectives: To design predictive models for the diagnosis of BL allergy, based on the clinical history of patients with suspicions of allergic reactions to BL.

Methods: The study included a retrospective phase in which records of patients consulting and explored for a suspicion of BL allergy (in the Allergy Unit of the University Hospital of Montpellier between September 1996 and September 2012) where used to construct predictive models; a prospective phase, in which we performed an external validation of the chosen models, in patients with suspicion of BL allergy recruited from 3 allergy centres (Montpellier, Nîmes, Narbonne), between March and November 2013. Data related to clinical history and allergy work-up results were retrieved and analysed. Logistic regression and decision tree method were used to design two models to predict the diagnosis of allergy to BL.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in consultation in allergology department for suspicion of allergy to beta lactamines

Exclusion Criteria:

* patient refusal to take part in the study
* pregnancy
* breast feeding women
* contraindication to provocation test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen in consultation in allergology department for suspicion of allergy to beta lactamines
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Provocation test | 18 months
  Results of provocation test for allergy diagnosis

SECONDARY OUTCOMES:
Questionnaire SF36 | 18 months
  Questionnaire SF36 will be compared to provocation test results
Questionnaire ENDA | 18 months
  Questionnaire ENDA will be compared to provocation test results

IPD SHARING:
Plan to Share IPD: No